CLINICAL TRIAL: NCT02447289
Title: Efficacy, Safety and Cost-effectiveness of Intranasal Sedation With Ketamine and Midazolam in Pediatric Dentistry: a Randomized Clinical Trial
Brief Title: Midazolam and Ketamine Effect Administered Through the Nose for Sedation of Children for Dental Treatment
Acronym: NASO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Luciane Ribeiro de Rezende Sucasas da Costa, Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 041530
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Child Behavior; Dental Caries
Keywords: Dental caries; Moderate sedation
MeSH Terms: conditions — Child Behavior; Dental Caries | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental (Experimental): Intranasal administration of ketamine (4.0 mg/kg, max. 100 mg) and midazolam (0.2 mg/kg, max. 5 mg)
  Interventions: Drug: Intranasal ketamine; Drug: Intranasal midazolam
- Comparator (Active Comparator): Oral administration of ketamine (4.0 mg/kg, max. 100 mg) and midazolam (0.5 mg/kg, max. 20 mg)
  Interventions: Drug: Oral ketamine; Drug: Oral midazolam
- Control (Active Comparator): Oral administration of midazolam (1.0 mg/kg, max. 20 mg)
  Interventions: Drug: Oral midazolam

INTERVENTIONS:
Drug: Intranasal ketamine — Ketamine injectable solution in a concentration of 50.0 mg/mL administered into the nose with an atomizer; dose of 4.0 mg/kg, maximum 100.0 mg
  Other Names: Ketamin S, Cristalia, São Paulo, Brazil
  Arms: Experimental
Drug: Oral ketamine — Ketamine injectable solution in a concentration of 50.0 mg/mL via oral route; dose of 4.0 mg/kg maximum 100.0 mg
  Other Names: Ketamin S, Cristalia, São Paulo, Brazil
  Arms: Comparator
Drug: Intranasal midazolam — Midazolam injectable solution in a concentration of 5.0 mg/mL administered into the nose with an atomizer; dose of 0.2 mg/kg, maximum 5.0 mg
  Other Names: Dormire injectable solution, Cristalia, São Paulo, Brazil
  Arms: Experimental
Drug: Oral midazolam — Midazolam oral solution in a concentration of 2.0 mg/mL via oral route; dose of 0.5 mg/kg, maximum 5.0 mg when associated with ketamine; dose of 1.0 mg/kg, maximum 20.0 mg when give as a solely agent
  Other Names: Dormire oral solution, Cristalia, São Paulo, Brazil
  Arms: Comparator; Control

SUMMARY:
Randomised clinical trial to test the efficacy, safety and cost-effectiveness of sedatives; masked, controlled, parallel design with three arms, phase 4.

DETAILED DESCRIPTION:
About 10% of children may have behavioral problems during dental treatment, but the evidence for sedative protocols that benefit the care in pediatric dentistry are still weak. This randomized, masked, controlled, parallel design study aims to evaluate the efficacy, safety and cost-effectiveness of intranasal sedation with ketamine / midazolam in healthy children aged 2 to 6 years old. Children will be selected among those with dental decay that do not allow dental treatment to be performed, and need at least two restorations under local anesthesia and rubber dam isolation. It is estimated a preliminarily a sample of 84 children equally divided into three groups: A) Ketamine (4.0 mg / kg up to 100 mg) + midazolam (0.2 mg / kg, maximum 5 mg) intranasally; B) ketamine (4.0 mg / kg up to 100 mg) + midazolam (0.5 mg / kg, maximum 20 mg) orally; C) midazolam (1.0 mg / kg, maximum 20 mg) orally. The hypothesis is that ketamine / midazolam combination, administered intranasally, it constitutes an effective sedative regime, safe and cost-effective for use in pediatric dentistry in the public service. The primary endpoint is the behavior of the child. Secondary endpoints are: sedative administration acceptance, procedure memory and salivary cortisol levels within each intervention group. Additionally, we will evaluate: the occurrence of pain and associated changes in facial expressions with potentially painful stimuli in children sedated for dental care; caregivers and paediatric dentists' stress and perception about sedation; adverse events that occur during and after administration of sedatives; cost-effectiveness of the sedative protocols. The experimental design is planned to minimize systematic and random errors and to contribute to higher level of evidence in future systematic reviews. The outcomes of this study have potential impact on public and private health practice, and may support institutional guidelines dealing with this theme.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I (healthy) or II (mild and controlled systemic disease such as persistent asthma)
* Small risk of airway obstruction (Mallampati less than 2 or tonsillar hypertrophy occupying less than 50% of the oropharynx)
* No medical history of neurological or cognitive changes
* Absence of facial deformities
* Term birth
* No use of drugs that may impair cognitive functions
* At least two teeth with cavities without pulp involvement, requiring dental restoration under local anesthesia and rubber dam

Exclusion Criteria:

* Positive or definitely positive behavior (Frankl et al, 1962) in a dental treatment session conducted by the research team

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-18 (Actual)

PRIMARY OUTCOMES:
Child's behavior measured by an observational scale | Participants will be followed for the duration of the dental session, an expected average of 40 minutes
  Children's behavior assessed by OSUBRS (Ohio State University Behavioral Rating Scale) in digital videos recorded during the administration. Scores: 1 - quiet, 2 - cry with movement, 3 - movement without cry; 4 - struggling. Satisfactory behavior means more than 60% of score 1 during the entire appointment.

SECONDARY OUTCOMES:
Acceptance of sedative administration measured by an observational scale | Participants will be assessed for the duration of the sedative administration, an expected average of 3 minutes
  Acceptance of the sedative administration, assessed by OSUBRS (Ohio State University Behavioral Rating Scale) minute by minute in digital videos recorded during the administration. Scores: 1 - quiet, 2 - cry with movement, 3 - movement without cry; 4 - struggling.
Participants' stress according to salivary cortisol | Change from baseline in the salivary cortisol at an expected average of 40 minutes
  Occurrence of stress during dental procedure, assessed by salivary cortisol in children, their accompanying parent and the dentist in charge; the ELISA test will determine changes in cortisol level during dental treatment
Pain measured by the FLACC Pain Assessment Tool | Participants will be followed in video files for the duration of the dental session, an expected average of 40 minutes
  Occurrence of pain and associated changes in body expressions with potentially painful stimuli in children sedated for dental care
Caregivers' and dentists' perceptions on sedation measured by a Visual Analogue Scale | During and soon after the dental session
  Perception of caregivers and dentists on sedation, through self-report
Child's perceptions on sedation through a semi-structured interview | One week after the dental session
  Child's perception concerning the dental treatment under sedation
Memory of the dental procedure at the immediate post-operative period measured by a validated test | Participants will be assessed for the recall of the dental procedure, at a time point of 20 minutes (average) after the end of the dental procedure
  Memory of the dental procedure, according to test with figures validated in Brazil. Amnesia will be reported if children do not recall the figures showed after sedative administration
Memory of the dental procedure after 24 hours measured by a validated test | Participants will be assessed for the recall of the dental procedure, at a time point of 24 hours (average) after the end of the dental procedure
  Memory of the dental procedure, according to test with figures validated in Brazil. Amnesia will be reported if children do not recall the figures showed after sedative administration
Adverse events during the dental procedure | Participants will be followed for the duration of the dental session, an expected average of 40 minutes
  Occurrence of adverse events assessed by the World SIVA tool; adverse events will be categorised into minor, sentinel and major
Post-operative adverse events | 24 hours
  Occurrence of adverse events while child is in the recovery room and after discharge, assessed by the World SIVA tool; adverse events will be categorised into minor, sentinel and major
Cost analysis | One year and a half
  Cost-effectiveness of different sedation protocols according to the methodology of health technologies assessment; the cost of each intervention will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Luciane R Costa, DDS, MS, PhD, Principal Investigator — Professor
Locations (1):
- Dental School, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be available as requested by the scientific journal where the manuscript is gonna be submitted

REFERENCES:
- [Derived] Sado-Filho J, Viana KA, Correa-Faria P, Costa LR, Costa PS. Randomized clinical trial on the efficacy of intranasal or oral ketamine-midazolam combinations compared to oral midazolam for outpatient pediatric sedation. PLoS One. 2019 Mar 11;14(3):e0213074. doi: 10.1371/journal.pone.0213074. eCollection 2019. PMID 30856181
- [Derived] Gomes HS, Miranda AR, Viana KA, Batista AC, Costa PS, Daher A, Machado GC, Sado-Filho J, Vieira LA, Correa-Faria P, Hosey MT, Costa LR. Intranasal sedation using ketamine and midazolam for pediatric dental treatment (NASO): study protocol for a randomized controlled trial. Trials. 2017 Apr 11;18(1):172. doi: 10.1186/s13063-017-1919-2. PMID 28399933